CLINICAL TRIAL: NCT00540540
Title: Measurements of Breast Tissue Optical Properties
Status: Withdrawn | Type: Observational
Why Stopped: According to NIH definition of clinical trial studies, this study does not meet requirement for clinical trial study.
Sponsor: University of California, Irvine (Other)
Collaborators: University of California, San Diego (Other); Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Bruce Tromberg, PhD, Director Beckman Laser Institute and Medical Clinic, Professor, Departments of Biomedical Engineering and Surgery, University of California, Irvine
Other Study IDs: 1995563
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Accessory; Breast Tissue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Diffuse Optical Spectroscopy — Breast properties scanning

SUMMARY:
Approximately twelve percent of the women in the United States will develop breast cancer, the most common form of cancer affecting women, with 183,000 new cases projected for 1995. Despite the increasing incidence, the age-adjusted death rate from carcinoma has remained relatively stable. Although the reason for this has not yet been demonstrated, this stability may be a direct consequence of early detection and improved therapy. Screening mammography as an early detection technique has been shown to reduce mortality by 23%. Mammographic abnormalities that go on to biopsy show 24% being positive for malignancy with great variability (6-75%). Breast biopsy is an expensive procedure with the risks of anesthesia and surgery which may be obviated by more specific non-invasive testing.

DETAILED DESCRIPTION:
Diffuse Optical Spectroscopic Imaging a new method for quantitative characterization of the optical properties of tissues. The diagnostic tools utilize anomalies in the transmission of diffusing near infra-red light for the rapid detection of oxygenated and deoxygenated hemoglobin, near infra-red absorbing drug levels, blood volume changes, and scattering properties in tissues.

Diffuse Optical Spectroscopic Imaging measurements of breast tissue optical properties probe is similar in shape to an ultrasound probe. The imaging can measurements on different areas of the breast including diseased location and normal area. Optical measurements can guided by co-registered ultrasound measurements for the purpose of determining lesion size and location. Each measurement will require about 5-60 seconds to record the data and calculate optical properties. The process will be repeated until an adequate number of measurements are performed and measurements take 30 to 90 minutes.

The researcher can determine that breast optical properties on demographic information, such as age and menopausal status as well as medical history.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant woman age 18 yrs and older.

Exclusion Criteria:

* pregnant woman and younger than 18 yrs of age.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will be selected from University of California Irvine Medical Clinic and Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 1995-12; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Healthy Breast | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bruce J Tromberg, Ph.D, Principal Investigator — Beckman Laser Institute
Locations (4):
- United States (4):
  - Pacific Breast Care Medical Clinic, Costa Mesa, California
  - Beckman Laser Institute University of California Irvine, Irvine, California
  - UCSD Regional Fertility Center, La Jolla San Diego, California
  - Chao Family Comprehensive Cancer Center, UCIMC, Orange, California